CLINICAL TRIAL: NCT00771589
Title: The Active Knee Prosthesis Will be Tested to Evaluate How Well it Improves the Gait Symmetry and Reduces the Metabolic Cost of an Amputee During Walking. The Prosthesis Will be Attached to the Socket of the Amputee.
Brief Title: Active Knee Prosthesis Study for Improvement of Locomotion for Above Knee Amputees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Hugh Herr, Ph.D., Massachusetts Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0804002682
Record Dates: First submitted 2008-10-08; First posted 2008-10-13 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prosthesis (Experimental): Motorized External Knee prosthesis for above knee amputees. Comprised of agonist and antagonist actuators to mimic behavior of knee joint during locomotion.
  Interventions: Device: Active Knee Prosthesis

INTERVENTIONS:
Device: Active Knee Prosthesis — Motorized External Knee Prosthesis for above knee amputees.
  Other Names: Agonist Antagonist Knee Prosthesis

SUMMARY:
The purpose of this study is to develop a robust, low-power, stable, and light weight, active knee prosthetic device that can dramatically increase gait symmetry and walking economy of a transfemoral amputee during walking.

State of the art prosthetic knees can be classified into three main classes: a) mechanically passive, b) variable-damping, and c) powered. Although the devices within each of these classes offer some advantages for above-knee amputees, their overall performance still presents some deficiencies. Artificial knees in the first two groups are predominantly damping devices, incapable of providing positive power output. Moreover, current powered prostheses are heavy and inefficient in their energy consumption, and/or they have a limited range of motion. To overcome such inadequacies, we have designed a novel prosthetic knee device with a biomimetic approach.

The design of the active knee prosthesis is inspired by the antagonistic muscle anatomy of the human knee joint. This device mimics the synergistic muscle activity at the knee using a double series-elastic actuator (SEA) system that resembles the major mono-articular muscle groups that help flex and extend the knee joint. The agonist-antagonist SEA knee architecture will allow for precise force control of the knee joint, mimicking the spring-like behavior of the human knee, as well as providing adequate energy for forward progression of the body. The SEA has been previously developed and tested on legged robots. Also, the SEA has been successfully applied to the development of an actuated ankle-foot orthoses (AAFO) at MIT AI Lab.

The mechanical architecture of the active knee prosthesis allows for independent engagement of flexion and extension tendon-like, series springs for the control of joint position and impedance, as well as net joint torque. Furthermore, this architecture permits a joint rotation with near zero friction, allowing the controller to take advantage of the passive dynamics of the system, thus, augmenting the overall energetic efficiency of the system.

DETAILED DESCRIPTION:
Healthy participants with above-knee amputations will be recruited. Participants will meet the following eligibility criteria. They will be experienced at prosthesis ambulation, with a capacity of ambulation at least at a K3 level (i.e. having the ability or potential for ambulation with variable cadence). Additionally, amputee participants will be generally healthy and will have no other musculoskeletal problems or any known cardiovascular, pulmonary or neurological disorders.

The research objective is to evaluate the efficacy of an active knee prosthesis that is designed to increase gait symmetry, speed, and to lower metabolic energy demands during walking.

For each amputee participant, a complete study will include three separate experimental sessions conducted in three different locations. These locations are: The Biomechatronics Group, MIT Media Laboratory; the Holodeck room in CSAIL at MIT; and the Indoor Track at MIT's Johnson Athletic Center. The time between experimental sessions will be approximately one to two weeks and the time duration of each session will be two to three hours. For each session, an amputee study participant will be asked to walk at slow, normal, and fast paces for two different conditions. The experimental conditions are:

1. Using an assigned commercially, available knee prosthesis (e.g. Otto Bock C-Leg or Ossur Rheo)
2. Using the active knee prosthesis

In the first session, each amputee participant will be scheduled to visit the Biomechatronics Group in The MIT Media Laboratory. The main purpose of this session is to qualitatively assess the degree to which the active prosthesis can improve amputee gait. Morphological data (for example, height, weight, limb length and circumference) of the participant will be recorded using the biomechanical data collection form. These data will be used during analysis of data gathered during the gait research sessions.

Each participant will be asked to walk along a 30-foot level walkway in the Biomechatronics Group. During the session, each participant will be asked to walk at slow, normal and fast paces for each of two walking conditions. For each condition and speed, approximately 10-15 trials will be performed. Parallel bars will be utilized to prevent any injury to the subject if he were to lose balance and fall. A safely harness attached to the ceiling will also be utilized if the subject makes that request. In addition, a member of the laboratory staff will also accompany the study participant to catch him in the event of a fall, if necessary. The participant may ask to rest or to terminate their participation in the study at any time.

Each participant will be walking on the platform 60-90 times for the entire first session, which should take approximately 2 hours. When using the active prosthesis with the walking program, our researchers will tune the parameters of the walking program to the participant's own gait pattern. The parameters used to tune the walking program will be recorded for use in Sessions 2 and 3.

In the second session, amputee study participants will be scheduled to visit the Holodeck room in CSAIL at MIT (Rm 33-339), that has installed the motion capture system to measure human movement. The main purpose of this session is to collect knee state, torque and power on amputees walking at slow, moderate and fast speeds. These active knee prosthetic data will then be compared to conventional prosthetic knee behaviors measured at the same three speeds.

Each participant will be asked to walk along a 30-foot level walkway in the Holodeck room in CSAIL at MIT. Before conducting experiments, one of the investigators will place reflective markers on the participant's skin with tape at specific points over joints of their body. These special markers are then seen by the cameras in the room (See Data Collection Instruments). During the session, each participant will be asked to walk at slow, normal and fast paces for each of two walking conditions. For each condition and speed, approximately 10-15 trials will be performed. Motion data is collected from cameras in the room and from the force plates that are placed in the walkway. As the device has been setup in the first session, two members of the laboratory staff will walk on each side of the participant throughout the experiment. The second session should take between 2 and 3 hours.

In the third session, each transfemoral amputee participant will be scheduled to visit the Indoor Track of the Johnson Athletic Center at MIT, which is located at the 2nd floor of the Athletic Center. The main purpose of this session is to test if the active knee prosthesis does, in fact, reduce the metabolic cost of amputee walking.

During the session, each participant will be asked to wear a Cosmed Oxygen Consumption (VO2) mask that will measure the metabolic rate. Two members of the laboratory staff will walk on each side of the participant throughout the experiment. The procedure for the experiment will be as follows:

The participant will be asked to wear the VO2 system and first walk for 8 minutes on the track with an assigned commercially, available above knee prosthesis (Otto Bock C-Leg or Ossur Rheo) to establish a control metabolic rate. After resting for 8 minutes, he/she will wear the active prosthesis and get acclimated to the device by walking for 5 minutes. He/she will then walk on the track for 8 minutes as we measure his/her metabolic rate with the device. The participant will then rest for another 8 minutes. This protocol will be repeated two additional times, and the entire experiment will take approximately 3 Hrs. Throughout the study, each participant will be videotaped and photographed to document the effect of the prosthesis on walking.

ELIGIBILITY:
Inclusion Criteria:

* They will be experienced at prosthesis ambulation
* Capacity of ambulation at least at a K3 level (i.e. having the ability or potential for ambulation with variable cadence).

Exclusion Criteria:

* Amputee participants will be generally healthy and will have no other musculoskeletal problems or any known cardiovascular, pulmonary or neurological disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-01 (Estimated); Study Completion 2009-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Herr, Ph.D., Principal Investigator — Massachusetts Institute of Technology
Locations (2):
- United States (2):
  - Biomechatronics Research Group, MIT, Cambridge, Massachusetts
  - LIfestyle Prosthetics & Orthotics, North Andover, Massachusetts

REFERENCES:
- [Derived] Martinez-Villalpando EC, Herr H. Agonist-antagonist active knee prosthesis: a preliminary study in level-ground walking. J Rehabil Res Dev. 2009;46(3):361-73. PMID 19675988